CLINICAL TRIAL: NCT00517257
Title: Atorvastatin Toronto Retinal Vein Occlusion Study (ATORVO)
Brief Title: Atorvastatin for the Treatment of Retinal Vein Occlusion
Acronym: ATORVO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other); Pfizer (Industry); Canadian Heart Research Centre (Other); Ontario Association of Optometrists (Other); Toronto Ophthalmological Society (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRA2580025
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Retinal Vein Occlusion; Retinal Vein Thrombosis; Central Retinal Vein Occlusion; Branch Retinal Vein Occlusion; Thrombosis
Keywords: Retinal vein occlusion; Retinal vein thrombosis; Central retinal vein occlusion; Branch retinal vein occlusion; Visual loss; Atorvastatin; Statin; Neovascularization; Thrombosis
MeSH Terms: conditions — Retinal Vein Occlusion; Thrombosis; Vision Disorders; Neovascularization, Pathologic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Atorvastatin 80 mg orally once daily for 24 weeks
  Interventions: Drug: Atorvastatin
- P (Placebo Comparator): Placebo tablet orally once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg orally once daily for 24 weeks
  Other Names: Lipitor
  Arms: A
Drug: Placebo — Placebo tablet orally once daily for 24 weeks
  Arms: P

SUMMARY:
The ATORVO study is designed to determine whether atorvastatin (Lipitor) can improve vision, when compared to placebo

DETAILED DESCRIPTION:
Retinal vein occlusion (RVO), a common cause of visual loss in the Western world, is a disease whose etiology resembles that of classic atherosclerosis. A therapy that lowers the risk of arterial and venous thrombosis would seem to be a reasonable approach to managing this disease, for which there is currently no treatment.

ATORVO is a randomized double-masked clinical trial comparing a daily dose of 80 mg of atorvastatin to matched placebo in persons recently diagnosed with RVO. At 24 weeks after randomization, we will evaluate each participant's visual acuity and the presence of secondary complications related to RVO.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years and older
* Diagnosed with CRVO or BRVO
* Visual acuity of 20/40 or worse in the affected eye
* Onset of current symptoms of loss of vision within the past 60 days
* Ability to understand spoken English

Exclusion Criteria:

* Current use of a statin or fibrate medication
* Known cardiovascular disease or revascularization, including coronary artery disease (myocardial infarction or angina), stroke or peripheral artery occlusion
* Known diabetes mellitus
* Known liver disease
* Serum low-density lipoprotein cholesterol (LDL-C) > 5.0 mmol/L
* Baseline serum triglycerides > 6.0 mmol/L
* Serum ALT above 115 U/L (i.e., 2.5 x upper limit of normal)
* Baseline serum creatinine > 250 µmol/L
* Ocular surgery within the past 90 days
* Planned ocular or cataract surgery within the study period
* Known retinal disease: age-related macular degeneration, retinal detachment or macular hole, or past history of vein occlusion
* Women who are pregnant or who are breastfeeding
* Participation in another clinical trial concurrently or within 30 days prior to screening
* Known allergy to fluorescein dye
* Current use of cyclosporine medication.
* Current use of an HIV protease inhibitor medication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-08; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Difference in improvement of at least 15 letters (3 lines) in Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity in the affected eye at 24 weeks in patients on active treatment vs. placebo. | 24 weeks

SECONDARY OUTCOMES:
Prevention of ocular neovascularization or need for laser treatment by 24 weeks. | 24 weeks
Reduction in macular edema, measured by optical coherence tomography at 24 weeks. | 24 weeks
Mean change in The National Eye Institute 25-Item Visual Function Questionnaire-25 (VFQ-25) score from 0 to 24 weeks. | 24 weeks
Composite of non-fatal myocardial infarction, hospitalization for acute coronary syndrome, receipt of coronary revascularization, stroke or death, by 52 weeks. | 24 weeks
Mean change in the concentration of serum total cholesterol, LDL-cholesterol and highly sensitive C-reactive protein at 0 and 24 weeks. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel G Ray, MD MSc, Principal Investigator — St. Michael's Hospital, University of Toronto; David Wong, MD, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada